CLINICAL TRIAL: NCT03039556
Title: The Influence of Acute Physical Inactivity on Metabolic Function in Older Men and Women
Brief Title: Step-reduction in Older Men and Women
Acronym: CDA-SR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Diabetes Association (Other)
Responsible Party: Principal Investigator, Stuart Phillips, Professor, McMaster University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0574
Record Dates: First submitted 2017-01-13; First posted 2017-02-01 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Older Adults; Reduced Physical Activity

ARMS (1):
- Change in physical activity for older adults (Experimental): Older adult participants undergo alterations in daily ambulation by completing Normal Daily Steps for one week, followed by a two-week Step-Reduction and a subsequent Return to Normal Daily Steps for two weeks
  Interventions: Behavioral: Normal Daily Steps; Behavioral: Step-Reduction; Behavioral: Return to Normal Daily Steps

INTERVENTIONS:
Behavioral: Normal Daily Steps — Complete normal daily ambulation for one week
Behavioral: Step-Reduction — Reduce daily ambulation to fewer than 1000 steps per day for two weeks
Behavioral: Return to Normal Daily Steps — Increase daily ambulation to 100% of normal daily step-count for two weeks

SUMMARY:
This study investigates the effects of two weeks of reduced daily ambulation and a subsequent return to normal physical activity on metabolic health of older adults.

DETAILED DESCRIPTION:
Aging results in a progressive loss of muscle mass that is accelerated by periods of muscular disuse, common for older adults during hospitalization or convalescence from illness. Transient physical inactivity has been shown to cause muscular atrophy and impairments in insulin sensitivity in both younger and older adults. However, the recovery capacity of older adults after such physical inactivity remains unknown. This study aims to determine the impact of two weeks of daily step reduction to ≤1000 steps per day, an experimental model mimicking short-term physical inactivity, on glycemic control in older adults and further investigate whether older adults are able to recover from the consequences of this inactivity simply by returning to their habitual activity for 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoker

Exclusion Criteria:

* Use of assistive walking devices
* Chronic use of analgesic or anti-inflammatory drugs
* History of neuromuscular problems or muscle and/or bone wasting disease
* Acute or chronic illness including cardiac, pulmonary, liver or kidney abnormalities, uncontrolled hypertension, insulin or non-insulin dependent diabetes or other metabolic disorders
* Daily use of statins, particularly simvastatin and atorvastatin
* Use of medications known to affect protein metabolism
* Normally complete fewer than 3000 steps per day

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change in Insulin Sensitivity | Measured at the end of each behavioural intervention (Week 1, Week 3, Week 5)
  Assessed via Matsuda ISI

SECONDARY OUTCOMES:
Change in lean tissue mass | Measured at the end of each behavioural intervention (Week 1, Week 3, Week 5)
  Assessed via Dual Energy X-Ray Absorptiometry
Change in Peak Isometric Maximal Voluntary Leg Extension Strength | Measured at the end of each behavioural intervention (Week 1, Week 3, Week 5)
  Assessed via muscle dynamometry
Change in Muscle Protein Synthesis | Measured at the end of each behavioural intervention (Week 1, Week 3, Week 5)
  Obtained via vastus lateralis muscle biopsy

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise Metabolism Research Laboratory, McMaster Univeristy, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Breen L, Stokes KA, Churchward-Venne TA, Moore DR, Baker SK, Smith K, Atherton PJ, Phillips SM. Two weeks of reduced activity decreases leg lean mass and induces "anabolic resistance" of myofibrillar protein synthesis in healthy elderly. J Clin Endocrinol Metab. 2013 Jun;98(6):2604-12. doi: 10.1210/jc.2013-1502. Epub 2013 Apr 15. PMID 23589526
- [Background] Devries MC, Breen L, Von Allmen M, MacDonald MJ, Moore DR, Offord EA, Horcajada MN, Breuille D, Phillips SM. Low-load resistance training during step-reduction attenuates declines in muscle mass and strength and enhances anabolic sensitivity in older men. Physiol Rep. 2015 Aug;3(8):e12493. doi: 10.14814/phy2.12493. PMID 26265753
- [Derived] McGlory C, von Allmen MT, Stokes T, Morton RW, Hector AJ, Lago BA, Raphenya AR, Smith BK, McArthur AG, Steinberg GR, Baker SK, Phillips SM. Failed Recovery of Glycemic Control and Myofibrillar Protein Synthesis With 2 wk of Physical Inactivity in Overweight, Prediabetic Older Adults. J Gerontol A Biol Sci Med Sci. 2018 Jul 9;73(8):1070-1077. doi: 10.1093/gerona/glx203. PMID 29095970